CLINICAL TRIAL: NCT05001165
Title: Dashboard Activated Services and Tele-Health for Heart Failure
Acronym: DASH-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Boback Ziaeian, Staff Cardiologist, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-000311
Record Dates: First submitted 2021-06-30; First posted 2021-08-11 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: heart failure; proactive outpatient management; learning health system; panel management; medical optimization
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients with perceived gaps in performance measures for guideline-directed medical therapies for heart failure with reduced ejection fraction will be chart-reviewed and called impromptu to receive point of care medication titration or reintegration into routine heart failure clinic. Patients lost to follow-up may be better identified using the HFrEF panel management tools.
  Interventions: Other: Proactive Panel Management Clinics for HFrEF
- Usual Care (No Intervention): A control group of patients with HFrEF will receive routine primary and cardiology care as currently indicated in routine scheduled clinic grids. Patients are at the discretion of their primary care and cardiology clinicians regarding whether further HFrEF optimization is warranted. While panel management data is available to all clinicians, clinical workflows and responsibilities do not encourage the use of panel data or response to performance measurement for HFrEF.

INTERVENTIONS:
Other: Proactive Panel Management Clinics for HFrEF — Novel clinic based on review of panel HFrEF data and impromptu telephone or video patient contacts/visits.
  Arms: Intervention

SUMMARY:
The Dashboard Activated Services and tele-Health for Heart Failure (DASH-HF) study is a pragmatic randomized controlled trial of a quality improvement (QI) intervention of a prospective panel management intervention to optimize medical treatment for Veterans with heart failure with reduced ejection fraction (HFrEF) compared to the receipt of usual VA health care services over a 6-month period of observation. The study will incorporate the existing VA Academic Detailing Heart Failure Dashboard (ADHFD) to target actionable patients with gaps in performance measures for guideline-directed medical therapies (GDMT). Patients with HFrEF are optimally managed by cardiovascular specialty clinics. Typically, patients are referred to cardiology or heart failure (HF) clinics from primary care, emergency department, or post-hospitalization clinicians and scheduled into clinic grids. These patients may be lost to follow-up or clinicians may miss opportunities to optimize GDMT for HFrEF. GDMT includes Class I indicated medications from the following classes: beta blockers (BB), angiotensin-converting enzyme inhibitor (ACE), angiotensin II receptor blockers (ARB), angiotensin receptor neprilysin inhibitor (ARNI), mineralocorticoid receptor antagonist (MRA), sodium-glucose cotransporter-2 inhibitor (SGLT2i). The intervention is designed around a novel prospective panel management clinic led by clinicians or clinical pharmacists using impromptu patient telephone calls or electronic communications with existing responsible clinicians.

DETAILED DESCRIPTION:
This is a randomized, pragmatic QI study designed to evaluate the effectiveness of proactive panel management to close gaps in evidence-based care for patients with HFrEF. The investigators will use the VA's ADHFD to generate a list of actionable patients with HFrEF and left ventricular ejection fraction (LVEF) ≤ 35%. After identifying a cohort of HFrEF patients from the ADHFD, the investigators will randomize individual patients on the actionable list to usual VA care or a novel proactive panel management clinic. Clinicians will be trained on how to use the dashboard information to identify opportunities for optimization based on detailed chart review. The proactive panel management intervention will use clinicians to perform an electronic chart review and call patients impromptu at their discretion to evaluate HFrEF management and opportunities to optimize GDMT. Each panel management clinic is staffed by a single cardiovascular clinician or trainee with cardiology (PI) supervision. All patients will receive chart review or telehealth notes brought to the attention of primary care and cardiology clinicians. Patients randomized to the intervention will only receive one chart review during a half-day panel management clinic with follow-up of any laboratory results or diagnostic tests as required and referral to HF or general cardiology clinic as deemed appropriate. The control arm consists of the usual delivery of health services with routine scheduled appointments for primary care or cardiology.

Outcomes will be assessed at 6-months from the last patient to receive the intervention. The study is powered to detect superiority of the intervention compared to usual care in optimizing GDMT for HFrEF. Treatment assignment is based on 1:1 randomization using fixed blocks (size=6) to assure an equivalent number of patients randomized to the intervention and usual care. Patients are randomized after a list of 300 actionable patients are generated from the ADHFD. Study participant numbers will be assigned to the list of patients sorted by optimization scores in Excel. The supervising statistician (AA) will generate concealed randomization assignments by participant identification numbers. The randomization assignments will be merged with baseline study dataset and exported as password protected Excel and PDF documents. Study investigators will divide the intervention arm into lists of 10 to 15 per half-day clinic. Patients not receiving chart review or phone call attempts will be reassigned to future panel management clinics until all patients receive the intervention. Patients that did not answer phone calls will receive chart review notes for primary care and cardiology clinicians and not be reassigned to future panel management clinics.

Study participants do not require informed consent as determined by the VA IRB review. Patients will receive all accepted standards of care and medications approved by the Food and Drug Administration for HFrEF indications. The VA Subcommittee for Research and Safety found an absence of any declared research-laboratory-based biohazards and granted exemption from continued review. The study will evaluate the effectiveness of the QI intervention, telephone/telemedicine panel management clinics, to more rapidly implement evidence-based care for patients with HFrEF. Patients in the usual care arm will be unaware they are part of the control group for the RCT. Intervention patients nor study staff are blinded to usual care or intervention assignments. Patients that receive the intervention will be informed this is a pilot quality improvement effort with informal consent before proceeding to the clinical interventions. Intervention patients may refuse to participate after being contacted by phone in the intervention.

Study enrollment is based on the inclusion and exclusion criteria used to filter the ADHFD list. A list of actionable patients with HFrEF will be exported for randomization. The GDMT optimization score will be automated for each patient on the extracted list (Table 1). A sample of 300 patients will be selected with the lowest GDMT composite scores. Once the final sample of the study is determined, patients will be randomized to usual care or the intervention. Intervention patients will be divided into smaller lists of 10 to 15 patients. These smaller lists will be assigned to proactive panel management clinics. Clinicians staffing the intervention clinics will review ADHFD data, review the electronic health record (EHR) and decide whether to proceed to evaluate and recommend treatment over the phone to patients directly. If clinicians did not have sufficient time to review all patients on their clinic list, they will be redistributed to future intervention clinics. Intervention clinics will be held until each patient assigned the intervention has a chart review or attempted telephone contact. A failure to contact a patient will trigger a letter to a patient or electronic communication to their primary care or cardiology clinician.

Prior to each ADHFD telehealth clinic (half-day clinic lasting 4 to 4.5 hours), clinicians will be sent a secure email that will include a password-protected Excel document of 15 patients with exported clinical summary data from the ADHFD. Clinicians will be instructed to chart-review patients and decide if an opportunity exists to further optimize the receipt of GDMT. Clinicians will also be given a document providing guidance on the sequence of GDMT optimization based on latest guidelines and VA policies (Supplement S1 GDMT Guidance Document). If a patient does not qualify for further optimization (i.e. chart documentation of prior intolerance, patient preference), a short note in the electronic health record (EHR) will document the chart review and inform the primary care clinician that based on chart review, no opportunity currently exists but they may consider further GDMT titration in the future. If a patient appears to have an opportunity for further titration, the clinician is encouraged to call the patient to see if they are available to discuss their HF care. If the patient agrees, a telehealth visit will take place over phone or switch to video. A formal telehealth cardiology visit will occur at the time of care. If the patient is interested but does not have time for a visit, a brief telephone note will be placed and a request for a future cardiology clinic visit will be requested. If a formal telehealth visit occurs, clinicians will be asked to inquire about key details around medication titration (Supplement S2 Interview Guide). The data from chart review and interviews will be documented on a password-protected Excel document (Supplement S3 Clinician Documentation Form). Any medication addition or titration will have indicated laboratory labs ordered per usual care. Lastly, clinicians will also be asked to administer a short survey with each participant based on a template at the end of the call proactive phone call (Supplement S2 Interview guide). Primary care and regular cardiology clinicians will be notified of any changes in medication management in the EHR. The study's lead (BZ, AV) will be available by phone to answer questions or problems that arise during the clinic. Supervision of patient encounters by clinical pharmacists, medical trainees, or advanced practice nurse practitioners and study protocols will be BZ as the licensed and boarded general cardiologist.

ELIGIBILITY:
Inclusion Criteria:

* Facility: Greater Los Angeles, CA
* Division: West LA VAMC
* Patient is eighteen years of age or older
* Patients has a primary diagnosis of HFrEF (last documented LVEF ≤35% per ADHFD algorithms)
* Patient has an estimated GFR greater than or equal to 30 mL/min
* Patient has a last documented potassium less than 5
* Patient has a last documented systolic blood pressure over 90 mm Hg
* Patient lacks at least one active prescription of a beta-blocker, ACE/ARB/ARNI, MRA, or SGLT2i
* There are no upcoming heart failure or primary care appointments in the upcoming 2 weeks.

Exclusion Criteria:

● Patient is currently hospitalized at WLA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boback Ziaeian, MD PhD, Principal Investigator — VA Greater Los Angeles Healthcare System
Locations (1):
- VA West Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verma A, Fonarow GC, Hsu JJ, Jackevicius CA, Vaghaiwalla Mody F, Nguyen A, Amidi O, Goldberg S, Vetrivel R, Upparapalli D, Theodoropoulos K, Gregorio S, Chang DS, Bostrom K, Althouse AD, Ziaeian B. DASH-HF Study: A Pragmatic Quality Improvement Randomized Implementation Trial for Patients With Heart Failure With Reduced Ejection Fraction. Circ Heart Fail. 2023 Sep;16(9):e010278. doi: 10.1161/CIRCHEARTFAILURE.122.010278. Epub 2023 Jul 26. PMID 37494051
- [Derived] Verma A, Fonarow GC, Hsu JJ, Jackevicius CA, Mody FV, Amidi O, Goldberg S, Upparapalli D, Theodoropoulos K, Gregorio S, Chang DS, Bostrom K, Althouse AD, Ziaeian B. The design of the Dashboard Activated Services and Telehealth for Heart Failure (DASH-HF) study: A pragmatic quality improvement randomized implementation trial for patients with heart failure with reduced ejection fraction. Contemp Clin Trials. 2022 Sep;120:106895. doi: 10.1016/j.cct.2022.106895. Epub 2022 Aug 24. PMID 36028192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Included patients were those over the age of 18 years, with a primary diagnosis of HFrEF with a last documented left ventricular ejection fraction ≤35%, an estimated eGFR ≥30 mL/minuter, and optimization potential score (OPS) of less than or equal to 5 out of 10, and no general cardiology or HF appointments in the upcoming 2 weeks. Exclusion criteria included if the dashboard indicated that the patient was currently hospitalized at the GLA VA.
Groups:
- Proactive Telehealth-based Clinics: The intervention included telehealth-based clinics, or DASH-HF clinics, for the target population. The clinics were led by clinicians (board-certified cardiologist, advanced HF cardiologist, nurse practitioner, cardiology fellow, advanced HF fellows [2], internal medicine resident and clinical pharmacists [2]).
  Clinicians staffing the clinic were provided a list of 10 to 15 intervention patients and worked at their own pace. The clinicians reviewed dashboard data and EHR and decided whether to proceed with a telehealth encounter. If the clinician did not have sufficient time to review all patients assigned to that day's clinic, the remaining patients were redistributed to future clinics. Patients who did not answer phone calls received mailed patient letters to encourage cardiology follow-up. Patients that were not able to be contacted were not reassigned to future panel management clinics. DASH-HF clinics were held until all subjects assigned to the intervention group had a chart review or attempted telephone contact.
- Usual Care: Patients with the VA Greater Los Angeles that received primary care or cardiovascular care as routinely scheduled.
Period: Overall Study
Arm/Group | Proactive Telehealth-based Clinics | Usual Care
Started | 150 | 150
Completed | 150 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proactive Telehealth-based Clinics | Usual Care | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.1 (11.5) | 72.1 (10.6) | 71.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 148 | 148 | 296
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 49 | 43 | 92
  White | 74 | 82 | 156
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Optimization Potential Score
Description: Change in composite score created for reaching target doses of guideline-directed medical therapies for HFrEF compared between treatment arms at the end of the study. Optimization Potential Scores ranges from 0 (least optimized) to 10 (full-optimized).
Time Frame: 6-months after all patients receive the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proactive Telehealth-based Clinics | Usual Care
Number analyzed (Participants) | 150 | 150
score on a scale | 2.9 (2.1) | 2.6 (2.1)
Statistical Analysis 1: Comparison: Proactive Telehealth-based Clinics vs Usual Care; Test type: Superiority; Regression, Linear; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.1 to 0.7]

2. Secondary Outcome: Change in Number of Patient Receiving ACE/ARB/ARNI
Description: Number of patients that receive an active prescription for angiotensin-converting enzyme inhibitor (ACE), angiotensin II receptor blockers (ARB), or angiotensin receptor neprilysin inhibitor (ARNI) compared between treatment arms at the end of the study.
Time Frame: 6-months after all patients receive the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Telehealth-based Clinics | Usual Care
Number analyzed (Participants) | 150 | 150
Participants | 97 | 86
Statistical Analysis 1: Comparison: Proactive Telehealth-based Clinics vs Usual Care; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.84 to 2.14]

3. Secondary Outcome: Change in the Number of Patients Receiving Beta-blockers
Description: Number of patients that receive an active prescription for beta-blockers compared between treatment arms at the end of the study.
Time Frame: 6-months after all patients receive the intervention
Population: Entire study population
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Telehealth-based Clinics | Usual Care
Number analyzed (Participants) | 150 | 150
Participants | 109 | 107
Statistical Analysis 1: Comparison: Proactive Telehealth-based Clinics vs Usual Care; Test type: Superiority; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.64 to 1.76]

4. Secondary Outcome: Change in the Number of Patients Receiving MRA
Description: Number of patients that receive an active prescription for mineralocorticoid receptor antagonist (MRA) compared between treatment arms at the end of the study.
Time Frame: 6-months after all patients receive the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Telehealth-based Clinics | Usual Care
Number analyzed (Participants) | 150 | 150
Participants | 53 | 47
Statistical Analysis 1: Comparison: Proactive Telehealth-based Clinics vs Usual Care; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.73 to 1.93]

5. Secondary Outcome: Change in Number of Patients Receiving ARNI
Description: Number of patients that receive an active prescription for angiotensin receptor neprilysin inhibitor (ARNI) compared between treatment arms at the end of the study. .
Time Frame: 6-months after all patients receive the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Telehealth-based Clinics | Usual Care
Number analyzed (Participants) | 150 | 150
Participants | 35 | 31
Statistical Analysis 1: Comparison: Proactive Telehealth-based Clinics vs Usual Care; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.68 to 2.05]

6. Secondary Outcome: Change in Number of Patients Receiving SGLT2i
Description: Number of patients that receive an active prescription for sodium-glucose cotransporter-2 inhibitor (SGLT2i) compared between treatment arms at the end of the study. .
Time Frame: 6-months after all patients receive the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Telehealth-based Clinics | Usual Care
Number analyzed (Participants) | 150 | 150
Participants | 44 | 33
Statistical Analysis 1: Comparison: Proactive Telehealth-based Clinics vs Usual Care; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.88 to 2.51]

7. Secondary Outcome: Total Number of Hospitalizations
Description: Total number of any cause hospitalizations compared between treatment arms at the end of the study.
Time Frame: 6-months
Measure: Number; unit: hospitalizations
Arm/Group | Proactive Telehealth-based Clinics | Usual Care
Number analyzed (Participants) | 150 | 150
hospitalizations | 29 | 17
Statistical Analysis 1: Comparison: Proactive Telehealth-based Clinics vs Usual Care; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 1.87, 95% CI 2-sided [0.99 to 3.64]

8. Secondary Outcome: Change in Total Deaths
Description: Total number of all-cause deaths compared between treatment arms at the end of the study.
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Telehealth-based Clinics | Usual Care
Number analyzed (Participants) | 150 | 150
Participants | 17 | 24
Statistical Analysis 1: Comparison: Proactive Telehealth-based Clinics vs Usual Care; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.34 to 1.33]

9. Other Pre Specified Outcome: Qualitative Analysis of Patient Satisfaction
Description: For only patients that received the intervention, we perform an informal survey of patient feelings about the telehealth intervention scaled from a range of 0 to 10 for satisfaction at the end of the visit. Zero represents no satisfaction with the intervention and 10 being complete satisfaction with the intervention.
  Control patients do not receive a survey question, since they did not receive the intervention.
Time Frame: At the end of the successful telehealth intervention. On average within one month of randomization.
Population: Patients Contacted
Measure: Mean (Standard Deviation); unit: Satisification Score (0-10)
Groups:
- Intervention Clinics: Half-day clinics that lasted three and half hours
Arm/Group | Intervention Clinics
Number analyzed (Participants) | 40
Satisification Score (0-10) | 9.3 (2.22)

10. Other Pre Specified Outcome: Average Number of Patients Contacted Per Half-day Clinic
Description: Average number of patients reviewed or contacted per half-day clinic to understand health services efficiency
Time Frame: After intervention is delivered (post-baseline) - on average within 1 month of randomization.
Population: Half-day clinics
Measure: Mean (Standard Deviation); unit: number of participants
Units Other Than Participants: Clinics
Arm/Group | Intervention Clinics
Number analyzed (Participants) | 150
Number analyzed (Clinics) | 21
number of participants | 7.14 (2.46)

11. Other Pre Specified Outcome: Clinician Time Per Patient
Description: This is estimated only for the intervention arm. Control patients did not receive the intervention so no time was spent per patient to compare. Clinician time spent per patient from opening chart to end of patient-specific intervention and documentation.
Time Frame: After intervention delivery (post-baseline). Within 1 month of the intervention on average.
Population: Patients chart reviewed
Measure: Mean (Standard Deviation); unit: Minutes spent per patient
Arm/Group | Intervention Clinics
Number analyzed (Participants) | 150
Minutes spent per patient | 33.72 (14.59)

12. Other Pre Specified Outcome: Average Number of Orders Placed Per Clinic
Description: 1. Average medication adjustments (stop, start, titration) per half-day clinic
  2. Average laboratory tests ordered per half-day clinic
  3. Average imaging/diagnostic procedures ordered per half-day clinic
  4. Average of referrals for consults/device therapy per half-day clinic
Time Frame: After intervention clinic delivered - on average within one month of randomization.
Population: Intervention group
Measure: Mean (Standard Deviation); unit: Number of orders
Units Other Than Participants: Clinics
Arm/Group | Intervention Clinics
Number analyzed (Participants) | 150
Number analyzed (Clinics) | 21
Number of orders
  Medication orders | 0.62 (1.07)
  Laboratory test orders | 0.81 (1.12)
  Imaging/diagnostic procedure orders | 0.57 (0.87)
  Referral for consult/device therapy orders | 0.76 (0.94)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Proactive Telehealth-based Clinics | Usual Care
All-Cause Mortality (participants affected / at risk) | 17/150 | 24/150
Serious Adverse Events (participants affected / at risk) | 43/150 | 38/150
Other Adverse Events (participants affected / at risk) | 0/150 | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proactive Telehealth-based Clinics (N=150) | Usual Care (N=150)
Hospitalizations (General disorders) | 29 (29) | 17 (17)
Mortality (General disorders) | 17 (17) | 24 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT05001165/Prot_001.pdf
  • Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT05001165/SAP_000.pdf